CLINICAL TRIAL: NCT02379156
Title: Thermoregulation and Cognition During Cool Ambient Exposure in Tetraplegia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, John Handrakis, PT, DPT, EdD, Research Health Science Specialist, James J. Peters Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HAN-14-045; 315696 (Other Grant/Funding Number: Craig H. Neilsen Foundation); 01589 (Other: JJPVAMC IRB)
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Tetraplegia; Hypothermia; Mild Cognitive Impairment
Keywords: Quadriplegia; Spinal Cord Injury; Body Temperature Regulation; Mild Cognitive Impairment
MeSH Terms: conditions — Quadriplegia; Hypothermia; Cognitive Dysfunction; Spinal Cord Injuries | interventions — Midodrine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Able-bodied Control Cool Temperature Exposure / No Drug (Other): Subjects are able-bodied (AB) persons, ages 18-65. AB participants were matched to the SCI group by age and gender. Procedure is exposure to cool temperature (64° F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance (Visit 1).
  Interventions: Other: Cool Temperature
- SCI Cool Temperature Exposure / No Drug (Experimental): Subjects are persons with tetraplegia: spinal cord lesion level C3 to T1, American Spinal Injury Association Impairment Scale (AIS) levels A and B, ages 18-65 years. Procedure is exposure to cool temperature (64° F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance (Visit 1).
  Interventions: Other: Cool Temperature
- SCI Cool Temperature Exposure with Drug (Experimental): Subjects are persons with tetraplegia who completed Visit 1 (no drug). Subjects are administered a 10 mg tablet of midodrine hydrochloride by a physician before being exposed to cool temperature (64° F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance (Visit 2).
  Interventions: Drug: Midodrine Hydrochloride; Other: Cool Temperature

INTERVENTIONS:
Drug: Midodrine Hydrochloride — Midodrine hydrochloride is an approved medication used to treat low blood pressure. We are using a standard dose of 10 mg (tablet) only one time to determine if the vascular-constricting effects of this drug will help keep warm blood closer to the body's core and improve the ability to maintain Tcore in a cool environment (off-label use). A physician will administer the drug once before the cool thermal challenge in subjects with tetraplegia only (Visit 2).
  Other Names: Gutron; ProAmatine; Amatine; Orvaten; Midodrine hydrochloride 10 mg tablet
  Arms: SCI Cool Temperature Exposure with Drug
Other: Cool Temperature — Subjects will be exposed to a routinely encountered cool temperature (64° F) for up to to 2 hours depending on the vital signs (BP, HR, Tcore) and tolerance (comfort).
  Other Names: 64° F

SUMMARY:
The ability to maintain normal core body temperature (Tcore = 98.6°F) is impaired in persons with a cervical spinal cord injury (tetraplegia). Despite the known deficits in the ability of persons with spinal cord injury (SCI) to maintain Tcore, and the effects of hypothermia to impair mental function in able-bodied (AB) persons, there has been no work to date addressing these issues in persons with tetraplegia.

Primary Aim: To determine if exposure of up to 2 hours to cool temperatures (64°F) causes Tcore to decrease in persons with tetraplegia, and if that decrease is associated with a decrease in cognitive function.

Primary Hypotheses: Based on our pilot data: (1) 66% of persons with tetraplegia and none of the matched controls will demonstrate a decline of 1.8°F in Tcore; (2) 80% of persons with tetraplegia and 30% of controls will have a decline of at least one T-score in Stroop Interference scores (a measure of executive function).

Secondary Aim: To determine the change in: (1) distal skin temperature, (2) metabolic rate, and (3) thermal sensitivity.

Secondary Hypothesis: Persons with tetraplegia will have less of a percent change in average distal skin temperatures and metabolic rate, and report lower thermal sensitivity ratings compared with AB controls.

Tertiary Aim: To determine if a 10 mg dose of an approved blood pressure-raising medicine (midodrine hydrochloride) will (1) reduce the decrease in Tcore and (2) prevent or delay the decline in cognitive performance in the group with tetraplegia compared to the exact same procedures performed on the day with no medicine (Visit 1) in that same group.

Tertiary Hypothesis: Through administering a one-time dose of midodrine, the medicine-induced decreased blood flow to the skin will lessen the decline in Tcore and prevent or delay the associated decline in cognitive performance compared to the changes in Tcore and cognitive performance during cool temperature exposure without midodrine in the same group with tetraplegia.

DETAILED DESCRIPTION:
This study will investigate the mechanisms contributing to thermoregulatory fragility in persons with tetraplegia when exposed to cool ambient temperatures that are routinely encountered during their activities of daily living (ADL). Subnormal body core temperatures and vulnerability to hypothermia (Tcore<95°F) have been reported in Veterans with tetraplegia upon exposure to relatively mild environmental temperatures. The impact that a drift in Tcore will be expected to have on cognitive performance, specifically working memory and executive function, will be demonstrated. These 2 areas of cognitive performance are vital for the ability to optimally care for one's self, which persons with higher cord lesions must excel at to ensure health and to attain the maximal degree of independence possible. The one-time administration of an alpha agonist, midodrine hydrochloride, in an attempt to attenuate the drift in Tcore and prevent or delay the expected decline in cognitive performance to exposure to cool on cognitive function will be investigated as well.

Preparation for Study Visits:

The study visits will be at least 1 day apart but no more than 2 weeks apart. Subjects will be provided a light, standard meal which they will be asked to eat 2 hours prior to their scheduled visit time. The meal will be either a plain bagel or 2 pieces of toast. For each visit, subjects will be asked to empty their bladders before their arrival and again upon arrival, if needed. Subjects will be asked to avoid caffeinated and alcoholic beverages and heavy exertion for 24-hours before testing. Subjects will wear minimal clothing (gym shorts, sports bra) during the study to maximize bare skin exposure to the cool temperature.

Visit 1: Cold Ambient Challenge Instrumentation: During the subject's first visit, a thin flexible rectal sensor will be placed 4 inches beyond the anal sphincter for Tcore measurement, and skin thermal sensors will be taped at 15 sites above and below the level of lesion for collection of skin temperature (Tsk). A mask will be placed over the subject's nose and mouth for measurement of exhaled gases from which resting metabolic rate will be calculated from analysis of expired gases (VO2) by a metabolic cart. Laser Doppler flowmetry (LDF) will be used to measure changes in microvascular perfusion by taping a laser doppler probe on the skin in the area of the ulnar styloid processes and medial malleoli bilaterally to confirm vasoconstriction. A pulse oximeter will be placed on the left second digit to obtain blood oxygen saturation and heart rate (HR). An automated blood pressure cuff will be placed above the right elbow to measure brachial blood pressure (BP). An intravenous catheter will be placed in the right antecubital or nearby vein and secured for sequential blood collection for blood hormones (cortisol and norepinephrine).

Baseline Collection: At the end of the 30-minute acclimation period (81°F), a 15-minute baseline (BL) collection of the following measures will be performed: Tcore, Tsk, and VO2 will be measured continuously; BP, HR, blood oxygenation, and thermal sensitivity will be measured at 5-minute intervals; 5 minutes of LDF will be measured at 10-minute intervals; a venous blood draw will be collected once for norepinephrine and cortisol concentrations. At the end of the BL period, a cognitive performance battery will be given.

Cool Ambient Challenge: Following the completion of the baseline period, subjects will be wheeled into a 64°F thermal room for 120 minutes or until Tcore ≤ 95°F. Tcore, Tsk, and VO2 will be continuously monitored for safety throughout the study, while BP, HR, blood oxygenation, and thermal sensitivity will be measured every 10 minutes. LDF will be measured for 5 minutes every 25 minutes, and venous blood will be collected every 60 minutes. The cognitive performance battery will be administered when Tcore has declined 1.8°F or is ≤ 95.9°F (in subjects with tetraplegia) or after 120 minutes of cold exposure (in both groups). A decrease in Tcore to ≤ 95°F, or moderate subject discomfort, will result in termination of the protocol. Subjects will be transferred to a warm room (81°F), covered with warming blankets, and given warm fluids. If symptoms continue, Dr. William Bauman will assess the subject and provide the appropriate care.

Visit 2: Cold Ambient Challenge with Midodrine Visit 2 will be completed in the subjects with tetraplegia who participated in Visit 1 and demonstrated an impaired ability to maintain Tcore. All procedures will be conducted in the seated position and will be the same as in Visit 1, with the exception of the oral administration of a 10 mg tablet of midodrine hydrochloride following the completion of the baseline period. Forty minutes after midodrine administration (in order for the medicine's effects to start), a second baseline collection will be performed and subjects will then be placed inside the 64°F thermal room for up to 2 hours or until Tcore ≤ 95°F. Data collection will follow the same schedule and be conducted in the same seated position as in Visit 1. During Visit 2, BP will be continuously monitored after midodrine administration for safety purposes. If subjects' BP increases to 160/90 mmHg, subjects will be seen by Dr. William Bauman, who may consider the administration of labetalol, if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Duration of SCI ≥1 year;
* Level of SCI C3-T1, AIS A & B;
* Age between 18 and 68 years.

Exclusion Criteria:

* Evidence of sympathetic integrity below the lesion level by the skin axon-reflex vasodilatation (SkARV) test;
* Known allergies to midodrine hydrochloride;
* Past Medical History (PMH) of diagnosed heart, kidney, peripheral vascular, or cerebral vascular disease, or diabetes mellitus;
* Hypertension (BP>140/90 mmHg);
* Untreated thyroid disease;
* Acute illness or infection;
* Current smoker;
* Pregnancy.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2021-07 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Handrakis, PT, DPT, EdD, Principal Investigator — James J. Peters VAMC
Locations (1):
- Center of Excellence for the Medical Consequences of SCI, James J Peters VAMC, The Bronx, New York, United States

REFERENCES:
- See also: Link to Research Center website. Look under Research tab to find Thermoregulation program. — http://www.scirc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Able-bodied Cool Temperature Exposure / No Drug: Subjects are able-bodied persons, ages 18-65 years matched for age and gender to the SCI group. Procedure is exposure to cool temperature (64° F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance (Visit 1).
  Cool Temperature: Subjects will be exposed to a routinely encountered cool temperature (64° F) for up to to 2 hours depending on the vital signs (Blood Pressure, Heart Rate, Tcore) and tolerance (comfort).
- SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine: The study consists of two visits separated by a 14-day washout period.
  The subjects are persons with tetraplegia: spinal cord lesion levels C3 to T1, American Spinal Injury Association Impairment Scale (AIS) levels A and B, ages 18-65. The Cool Temperature Exposure consists of a 64° F temperature-controlled room for up to 2 hours.
  Visit 1 (120 minutes, SCI Cool Exposure without drug) consists of SCI Cool Temperature Exposure for up to 2 hours to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance.
  A washout period of 14 days separates Visit 1 and Visit 2.
  In Visit 2 (120 minutes, SCI Cool Exposure with drug), subjects who completed Visit 1 and did not rescind their study participation during the washout period are administered a 10 mg tablet of midodrine hydrochloride by a physician before being exposed to cool temperature (64° F) for up to 2 hours in a temperature-controlled room to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance.
Period: Overall Study
Arm/Group | Able-bodied Cool Temperature Exposure / No Drug | SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine
Started | 15 | 15
Completed | 15 | 12 (Of the 15 participants with Spinal Cord Injury (SCI) who started the Cool Temperature/No Drug arm, only 14 completed Visit 1. One participant failed the screening. Furthermore, only 12 of the 14 participants who completed Visit 1 proceeded to Visit 2.)
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Population: The reported SCI baseline characteristics pertain to the 12 individuals that completed both Visit 1 and Visit 2.
Groups:
- SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine: The study consists of two visits separated by a 14-day washout period. The subjects are persons with tetraplegia: spinal cord lesion levels C3 to T1, AIS levels A and B, ages 18-65. The Cool Temperature Exposure consists of a 64° F temperature-controlled room for up to 2 hours.
  Visit 1 (120 minutes, SCI Cool Exposure without drug) consists of SCI Cool Temperature Exposure for up to 2 hours to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance.
  A washout period of 14 days separates Visit 1 and Visit 2. In Visit 2 (120 minutes, SCI Cool Exposure with drug), subjects who completed Visit 1 and did not rescind their study participation during the washout period are administered a 10 mg tablet of midodrine hydrochloride by a physician before being exposed to cool temperature (64° F) for up to 2 hours in a temperature-controlled room to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance.
- Total: Total of all reporting groups
Arm/Group | Able-bodied Cool Temperature Exposure / No Drug | SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (11.38) | 37.1 (7.9) | 41.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 13 | 10 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Non-Hispanic | 3 | 5 | 8
  Race/Ethnicity: Black or African American | 9 | 0 | 9
  Race/Ethnicity: Hispanic | 2 | 7 | 9
  Race/Ethnicity: Asian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 12 | 27
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 26.42 (5.28) | 25.19 (2.77) | 25.93 (0.46)

OUTCOME MEASURES:

1. Primary Outcome: Change in Core Body Temperature
Description: We measured the effects of cool temperature (64°F) exposure, of up to 120 minutes, on the ability to maintain a constant Tcore (i.e., Tcore of 98.6°F) in all intervention arms.
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: °C
Groups:
- Able-bodied Control Cool Temperature Exposure / No Drug: Subjects are able-bodied (AB) persons, ages 18-65. AB participants were matched to the SCI group by age and gender. Procedure is exposure to cool temperature (64° F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance (Visit 1).
  Cool Temperature: Subjects will be exposed to a routinely encountered cool temperature (64° F) for up to to 2 hours depending on the vital signs (Blood Pressure (BP), Heart Rate (HR), Tcore) and tolerance (comfort).
Arm/Group | Able-bodied Control Cool Temperature Exposure / No Drug | SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine
Number analyzed (Participants) | 15 | 12
°C
  Change in Core Temperature during Cool Temperature Exposure (64 °F, 120 minutes), no drug | -0.24 (0.33) | -0.97 (0.33)
  Change in Core Temperature during Cool Temperature Exposure (64 °F, 120 minutes), drug | NA (NA) — Midodrine hydrochloride (HCl) was not given to Able-Bodied controls. | 0.79 (0.28)
Statistical Analysis 1: Comparison: Able-bodied Control Cool Temperature Exposure / No Drug; Between-group differences in the change in core body temperature (Tcore) from baseline (BL) values to after cold exposure (Cold) were analyzed using a Mixed Model ANOVA. We hypothesized that participants with tetraplegia would have a greater decrease in Tcore when exposed to cool ambient temperature than control participants exposed to the same cool ambient temperature; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine; Within-group differences in the change in (Tcore) in the participants with tetraplegia from BL values to Cold, with and without a dose of 10 mg of midodrine (two separate visits), were analyzed using a Repeated Measures ANOVA; Test type: Superiority; p = 0.006, ANOVA

2. Secondary Outcome: Percent Change in Cognitive Performance - Wechsler Adult Intelligence Scale 4th Edition (WAIS IV)
Description: Cognitive performance was assessed using the Wechsler Adult Intelligence Scale 4th Edition (WAIS-IV) Digit Span test, which measures working memory and attention. The test consists of three subtests: Digit Span Forward, Digit Span Backward, and Digit Span Sequencing. Each subtest yields a scaled score ranging from 1 to 19 based on age-based normative data. The total scaled score is obtained by summing the three subtest scores, resulting in a possible total scaled score range of 3 to 57.
  For each subtest (Digit Span Forward, Digit Span Backward, and Digit Span Sequencing) and for the total scaled score, higher scores indicate better working memory performance (better outcome), while lower scores indicate poorer working memory performance (worse outcome).
  Assessments were conducted at baseline (BL) and after cold ambient exposure. The reported results represent the percent change in each participant's total scaled score from baseline to post-exposure ([(Cold - BL) / BL] × 100).
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Able-bodied Cool Temperature Exposure / No Drug: Subjects are able-bodied persons, ages 18-65 years matched for age and gender to the SCI group. Procedure is exposure to cool temperature (64° F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance (Visit 1).
  Cool Temperature: Subjects will be exposed to a routinely encountered cool temperature (64° F) for up to to 2 hours depending on the vital signs (BP, HR, Tcore) and tolerance (comfort).
Arm/Group | Able-bodied Cool Temperature Exposure / No Drug | SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine
Number analyzed (Participants) | 15 | 12
Percent Change
  Percent Change in Cognitive performance - (WAIS IV), no drug | 3.81 (15.90) | -11.08 (21.47)
  Percent Change in Cognitive performance - (WAIS IV), drug | NA (NA) — Midodrine HCl was not given to Able-Bodied controls. | -1.73 (16.98)
Statistical Analysis 1: Comparison: Able-bodied Cool Temperature Exposure / No Drug; Between-group differences in the percent change in total WAIS IV scores from BL to after cold ambient exposure were analyzed using an independent samples T-test. We hypothesized that participants with tetraplegia would have a greater percent change in total WAIS IV scores due to impaired cognitive function post cool ambient exposure; Test type: Superiority; p = .042, t-test, 2 sided
Statistical Analysis 2: Comparison: SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine; Within-group differences in the percent change in total WAIS IV scores from BL to after cold ambient exposure were analyzed using a paired samples t-test. We hypothesized that participants with tetraplegia in the "No Drug" condition would have a greater percent change in total WAIS IV scores than the same participants in the "With drug" condition; Test type: Superiority; p = 0.149, t-test, 2 sided

3. Secondary Outcome: Change in Distal Skin Temperature (Tsk)
Description: We measured the effects of cool ambient exposure (64°F) in each intervention arm by taping 4 thermocouples to the skin of distal areas of the extremities (i.e. the fingers and toes).
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Able-bodied Control Cool Temperature Exposure / No Drug | SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine
Number analyzed (Participants) | 15 | 12
°C
  Change in Distal Skin Temperature (Tsk), no drug | -10.82 (2.10) | -4.35 (1.69)
  Change in Distal Skin Temperature (Tsk), drug | NA (NA) — Midodrine HCl was not given to Able-Bodied controls. | -1.45 (2.25)
Statistical Analysis 1: Comparison: Able-bodied Control Cool Temperature Exposure / No Drug; Between-group differences in the change in distal skin temperature temperature (Tsk) from baseline (BL) values to after ambient cold exposure (Cold) were analyzed using a mixed-model ANOVA for the AB vs Tetra comparison. We hypothesized that participants with tetraplegia would have a smaller change in Tsk due to being in a constant state of vasodilation; Test type: Superiority; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine; Within-group differences in the change in distal skin temperature temperature (Tsk) from baseline (BL) values to after ambient cold exposure (Cold) were analyzed using a repeated measures ANOVA for the within-group comparison of drug vs no drug in the tetraplegia group. We hypothesized that participants with tetraplegia with drug would have a larger decrease in Tsk due to enhanced peripheral vasoconstriction due to the drug's effects; Test type: Superiority; p < .001, ANOVA

4. Secondary Outcome: Percent Change in Microvascular Perfusion
Description: We measured the effects of ambient cool exposure (64°F), for up to 120 minutes, on microvascular perfusion by taping laser doppler flowmetry (LDF) probes to the skin of the hands and feet. LDF was measured in all intervention arms and compared the percent changes in microvascular perfusion within and between groups.
Time Frame: Up to 120 minutes
Measure: Mean (Standard Deviation); unit: Percent change in arbitrary units
Arm/Group | Able-bodied Control Cool Temperature Exposure / No Drug | SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine
Number analyzed (Participants) | 15 | 12
Percent change in arbitrary units
  Percent Change in Microvascular Perfusion, no drug | -56.13 (12.40) | -10.93 (41.34)
  Percent Change in Microvascular Perfusion, drug | NA (NA) — Midodrine HCl was not given to Able-Bodied controls. | -29.42 (10.90)
Statistical Analysis 1: Comparison: Able-bodied Control Cool Temperature Exposure / No Drug; Between-group differences in the percent change in microvascular perfusion from baseline to after cool ambient exposure were analyzed using independent samples T-test. We hypothesized that participants with tetraplegia would have a smaller percent change in microvascular perfusion due impaired vasomotor control which causes a constant state of vasodilation; Test type: Superiority; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine; Within-group differences in the percent change in microvascular perfusion from baseline to after cool ambient exposure were analyzed using a paired samples t-test. We hypothesized that participants with tetraplegia in the "No Drug" condition would have a smaller percent change in microvascular perfusion due impaired vasomotor control which causes a constant state of vasodilation; Test type: Superiority; p = 0.066, t-test, 2 sided

5. Secondary Outcome: Percent Change in Oxygen Consumption (VO2)
Description: We measured the effects of ambient cool exposure (64°F), for up to 120 minutes, on oxygen consumption (VO2) as a measure of resting metabolic rate. VO2 was measured in all intervention arms to compare the percent changes within and between groups.
Time Frame: Up to 120 minutes.
Measure: Mean (Standard Deviation); unit: percent change in VO2
Arm/Group | Able-bodied Control Cool Temperature Exposure / No Drug | SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine
Number analyzed (Participants) | 14 | 12
percent change in VO2
  Percent Change in oxygen consumption (VO2), no drug | -6.25 (11.36) | 1.88 (14.80)
  Percent Change in oxygen consumption (VO2), drug | NA (NA) — Midodrine HCl was not given to Able-Bodied controls. | 1.13 (16.72)
Statistical Analysis 1: Comparison: Able-bodied Control Cool Temperature Exposure / No Drug; Between-group differences in the percent change in VO2 from baseline to after cool ambient exposure were analyzed using independent samples t-test. We hypothesized that participants with tetraplegia would have a smaller percent change in VO2 consumption; Test type: Superiority; p = 0.127, t-test, 2 sided
Statistical Analysis 2: Comparison: SCI Cool Temperature Exposure With no Drug First, Then SCI Cool Temperature Exposure With Midodrine; Within-group differences in the percent change in VO2 consumption from baseline to after cool ambient exposure were analyzed using a paired samples t-test. We hypothesized that participants with tetraplegia in the "No Drug" condition would have a greater percent change in VO2 consumption due to impaired vasoconstriction and greater heat loss compared to the "With Drug" condition, in response to cool ambient exposure; Test type: Superiority; p = 0.964, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were reported within five business days to the VA's Institutional Review Board (IRB) via an Adverse Event form and were also included on the Adverse Events log on the annual continuing review application in accordance with VA IRB policy. Adverse event data were collected through study completion, up to 14 days.
Groups:
- Able-bodied Cool Temperature Exposure: Subjects are able-bodied persons, ages 18-65 years matched for age and gender to the SCI group. Procedure is exposure to cool temperature (64° F) for up to 2 hours in a temperature-controlled room in order to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance (Visit 1).
  Cool Temperature: Subjects will be exposed to a routinely encountered cool temperature (64° F) for up to to 2 hours depending on the vital signs (BP, HR, Tcore) and tolerance (comfort).
- SCI Cool Temperature Exposure: The study consists of two visits separated by a 14-day washout period.
  The subjects are persons with tetraplegia: spinal cord lesion levels C3 to T1, AIS levels A and B, ages 18-65. The Cool Temperature Exposure consists of a 64° F temperature-controlled room for up to 2 hours.
  Visit 1 (120 minutes, SCI Cool Temperature Exposure without drug) consists of SCI Cool Temperature Exposure for up to 2 hours to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance.
- SCI Cool Temperature Exposure With Midodrine: The study consists of two visits separated by a 14-day washout period.
  The subjects are persons with tetraplegia: spinal cord lesion levels C3 to T1, AIS levels A and B, ages 18-65. The Cool Temperature Exposure consists of a 64° F temperature-controlled room for up to 2 hours.
  In Visit 2 (120 minutes, SCI Cool Temperature Exposure With Midodrine), subjects who completed Visit 1 and did not rescind their study participation during the washout period are administered a 10 mg tablet of midodrine hydrochloride by a physician before being exposed to cool temperature (64° F) for up to 2 hours in a temperature-controlled room to assess the body's temperature-regulating mechanisms and any associated change in cognitive performance.
Arm/Group | Able-bodied Cool Temperature Exposure | SCI Cool Temperature Exposure | SCI Cool Temperature Exposure With Midodrine
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT02379156/Prot_SAP_000.pdf